CLINICAL TRIAL: NCT03046277
Title: Short- and Long-Term Renal Outcomes Following Lung Transplantation- A Single-Centre Experience
Brief Title: Short- and Long-Term Renal Outcomes Following Lung Transplantation
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior Physician Nephrology, University of Giessen
Other Study IDs: UGiessen
Record Dates: First submitted 2017-02-04; First posted 2017-02-08 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Lung Transplantation; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Collection of only residual material (blood, urine) was done for Deutsche Zentrum für Lungenforschung Biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing LTx: Retrospective analysis of clinical data
  Interventions: Other: No intervention
- Patients with pretransplant renal functional reserve testing: Prospective analysis of clinical data
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Evaluation of acute kidney injury, renal recovery and development of chronic kidney disease in patients undergoing lung transplantation

DETAILED DESCRIPTION:
It is well described that acute kidney injury and development of chronic kidney disease significantly impact short- and long-term survival after lung transplantation. However, there is limited data about prevalence of kidney disease according to current KDIGO consensus guidelines. It is the aim of this study to describe short- and long-term renal outcomes following lung transplantation. Selected patients who underwent prospective pretransplant renal functional reserve testing with high oral protein load will be analyzed separately in respect to occurrence of acute kidney injury following lung transplantation and development of chronic kidney disease.

ELIGIBILITY:
For retrospective analysis for all patients undergoing lung transplantation:

Inclusion Criteria:

* Older than 18 years

Exclusion Criteria:

* Patients with eGFR <15ml/min/1.73m2 or with chronic dialysis treatment prior LTx
* Patients undergoing retransplantation and multiorgan transplantation

For prospective study involving patients with pretransplant renal functional reserve testing

Exclusion criteria:

* as above
* unable to perform renal functional reserve testing (e.g., due to critical illness)
* pre-existing acute kidney injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing lung transplantation at University Hospital Giessen between 2003 and 2016. Subgroup of patients who underwent pretransplant renal functional reserve testing will be analyzed separately.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Impact of acute kidney injury (AKI) after lung transplantation on long-term renal function decline. | 7 days
  AKI defined by KDIGO consensus criteria

SECONDARY OUTCOMES:
Impact of sustained reversal versus non-recovery after AKI on long-term renal function decline after lung transplantation. | 3 years
  AKI and CKD defined by KDIGO consensus criteria
Risk factors associated with development of AKI and CKD after lung transplantation | 3 years
  AKI and CKD defined by KDIGO consensus criteria
Whether development of CKD is an independent risk factor for increased rejection rate and death after lung transplantation. | 3 years
  CKD defined by KDIGO consensus criteria
Association between pretransplant renal functional reserve with acute kidney injury after after lung transplantation. | 7 days
  AKI defined by KDIGO consensus criteria
Association between pretransplant renal functional reserve and renal function loss after lung transplantation. | 1 year
  24h-creatinine clearance, estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — University Hospital Giessen and Marburg, Giessen, Department of Internal Medicine II, Division of Pulmonology, Nephrology and Critical Care Medicine
Locations (1):
- University Clinic Giessen and Marburg - Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husain-Syed F, Ferrari F, Sharma A, Danesi TH, Bezerra P, Lopez-Giacoman S, Samoni S, de Cal M, Corradi V, Virzi GM, De Rosa S, Mucino Bermejo MJ, Estremadoyro C, Villa G, Zaragoza JJ, Caprara C, Brocca A, Birk HW, Walmrath HD, Seeger W, Nalesso F, Zanella M, Brendolan A, Giavarina D, Salvador L, Bellomo R, Rosner MH, Kellum JA, Ronco C. Preoperative Renal Functional Reserve Predicts Risk of Acute Kidney Injury After Cardiac Operation. Ann Thorac Surg. 2018 Apr;105(4):1094-1101. doi: 10.1016/j.athoracsur.2017.12.034. Epub 2018 Jan 31. PMID 29382510
- [Result] Fidalgo P, Ahmed M, Meyer SR, Lien D, Weinkauf J, Cardoso FS, Jackson K, Bagshaw SM. Incidence and outcomes of acute kidney injury following orthotopic lung transplantation: a population-based cohort study. Nephrol Dial Transplant. 2014 Sep;29(9):1702-9. doi: 10.1093/ndt/gfu226. Epub 2014 Jun 23. PMID 24957809
- [Result] Fidalgo P, Ahmed M, Meyer SR, Lien D, Weinkauf J, Kapasi A, Cardoso FS, Jackson K, Bagshaw SM. Association between transient acute kidney injury and morbidity and mortality after lung transplantation: a retrospective cohort study. J Crit Care. 2014 Dec;29(6):1028-34. doi: 10.1016/j.jcrc.2014.07.024. Epub 2014 Jul 31. PMID 25138690
- [Result] Canales M, Youssef P, Spong R, Ishani A, Savik K, Hertz M, Ibrahim HN. Predictors of chronic kidney disease in long-term survivors of lung and heart-lung transplantation. Am J Transplant. 2006 Sep;6(9):2157-63. doi: 10.1111/j.1600-6143.2006.01458.x. Epub 2006 Jul 6. PMID 16827787
- [Derived] Kuhnert S, Sommerlad J, Gall H, Weder MM, Wolff M, Eberle S, Sander M, Reichert M, Koch C, Askevold I, Hecker A, Padberg W, Ostermann M, Mehta R, Ronco C, Birk HW, Seeger W, Mayer K, Hecker M, Husain-Syed F. Postoperative Fluid Accumulation is Associated With Underestimation of AKI Severity in Lung Transplant Recipients. Clin Transplant. 2024 Sep;38(9):e15457. doi: 10.1111/ctr.15457. PMID 39282762